CLINICAL TRIAL: NCT03229317
Title: Respiratory Outcome According to Early Maternal Vitamin D Status During Pregnancy in Children Aged 5 to 6 Years Old
Brief Title: Respiratory Outcome of Children From the FEPED Cohort
Acronym: RESPIFEPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: K160907J; 2017-A01193-50 (Other: IDRCB)
Record Dates: First submitted 2017-07-03; First posted 2017-07-25 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Asthma in Children
Keywords: Lung function; Children; Vitamin D; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Plethysmography — Lung plethysmography

SUMMARY:
Early lung function deficits represent a significant risk factor for the evolution toward chronic obstructive pulmonary disease later in life. Prematurity and in utero tobacco smoke exposure are already known to predispose children to develop a non-reversible obstructive ventilatory defect in adulthood. The role of vitamin D status during pregnancy is less certain. In humans, low vitamin D concentrations during pregnancy are associated to an increased risk of asthma in children. In murine models, low vitamin D concentrations during pregnancy are associated to structural abnormalities of the airways in mouse pups. Investigators hypothesized that vitamin D play a role in early airways development, from the first trimester of pregnancy. To bring arguments to this hypothesis, the investigators will study the association of airway resistance in children aged 5 to 6 years old with the concentration of vitamin D during the first trimester of pregnancy in their mothers.

DETAILED DESCRIPTION:
Children aged 5 to 6 years old will be included from the FEPED cohort. The FEPED cohort is a cohort of French pregnant women designed to study the association between vitamin D status during pregnancy and the risk of pre-eclampsia. Vitamin D concentration at first and third trimester of pregnancy as well as in cord blood is available for 1400 women. Investigators will include 200 children born from these women. Children will undergo lung function tests and prick-tests and parents will answer the ISAAC questionnaire that is a standardised questionnaire designed to evaluate asthma and rhinitis symptoms. The main outcome of this study will be specific airway resistance. The investigators will look for an association between specific airway resistance and vitamin D concentration measured during the first trimester of pregnancy in their mothers.

ELIGIBILITY:
Inclusion Criteria:

* term-born child (gestational age ≥ 37 weeks of post-menstrual age) whose mother was included in the FEPED cohort
* measure of vitamin D concentration available at the first and third trimester of pregnancy and in cord blood
* cord blood sample available for DNA extraction
* child's age between 5 and 6 years old at the time of participation
* written informed consent obtained from the legal guardian of the child
* health insurance

Exclusion Criteria:

* parent's' refusal
* underlying disease that does not allow the performance of lung function tests

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: term-born child (gestational age ≥ 37 weeks of post-menstrual age) whose mother was included in the FEPED cohort, with measure of vitamin D concentration available at the first and third trimester of pregnancy and in cord blood
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Specific airway resistance measured by plethysmography | 1 day
  The measure of this outcome will be compared between children with a concentration of vitamin D during the first trimester of pregnancy < 20 ng/ml and children with a concentration ≥ 20 ng/ml

SECONDARY OUTCOMES:
Interrupter airway resistance measured by the interrupter technique using a pneumotachograph | 1 day
  This secondary outcome is another way to measure airway resistance. The measure of this outcome will be also compared between children with a concentration of vitamin D during the first trimester of pregnancy < 20 ng/ml and children with a concentration ≥ 20 ng/ml
Residual functional capacity measured by the helium dilution technique | 1 day
  This secondary outcome is another lung function parameter that will allow to evaluate lung volumes of the participants. The measure of this outcome will also be compared between children with a concentration of vitamin D during the first trimester of pregnancy < 20 ng/ml and children with a concentration ≥ 20 ng/ml
Occurrence of one wheezing episode | 1 day
Age of the first wheezing episode | 1 day
Occurrence of Asthma at age 3 years old | 1 day
Occurrence of Asthma at age 5 or 6 years old | 1 day
Allergenic sensitizations determined by skin prick-tests | 1 day
Genotype of 4 single nucleotide polymorphisms related to vitamin D metabolism | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Alice HADCHOUEL, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Alexandra BENACHI, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Armand Trousseau Hospital, Paris, Paris
  - Necker Enfants-malades Hospital, Paris, Paris
  - Robert Debré Hospital, Paris, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chawes BL, Bonnelykke K, Stokholm J, Vissing NH, Bjarnadottir E, Schoos AM, Wolsk HM, Pedersen TM, Vinding RK, Thorsteinsdottir S, Arianto L, Hallas HW, Heickendorff L, Brix S, Rasmussen MA, Bisgaard H. Effect of Vitamin D3 Supplementation During Pregnancy on Risk of Persistent Wheeze in the Offspring: A Randomized Clinical Trial. JAMA. 2016 Jan 26;315(4):353-61. doi: 10.1001/jama.2015.18318. PMID 26813208
- [Background] Litonjua AA, Carey VJ, Laranjo N, Harshfield BJ, McElrath TF, O'Connor GT, Sandel M, Iverson RE Jr, Lee-Paritz A, Strunk RC, Bacharier LB, Macones GA, Zeiger RS, Schatz M, Hollis BW, Hornsby E, Hawrylowicz C, Wu AC, Weiss ST. Effect of Prenatal Supplementation With Vitamin D on Asthma or Recurrent Wheezing in Offspring by Age 3 Years: The VDAART Randomized Clinical Trial. JAMA. 2016 Jan 26;315(4):362-70. doi: 10.1001/jama.2015.18589. PMID 26813209
- [Background] Wolsk HM, Harshfield BJ, Laranjo N, Carey VJ, O'Connor G, Sandel M, Strunk RC, Bacharier LB, Zeiger RS, Schatz M, Hollis BW, Weiss ST, Litonjua AA. Vitamin D supplementation in pregnancy, prenatal 25(OH)D levels, race, and subsequent asthma or recurrent wheeze in offspring: Secondary analyses from the Vitamin D Antenatal Asthma Reduction Trial. J Allergy Clin Immunol. 2017 Nov;140(5):1423-1429.e5. doi: 10.1016/j.jaci.2017.01.013. Epub 2017 Mar 9. PMID 28285844
- [Background] Gazibara T, den Dekker HT, de Jongste JC, McGrath JJ, Eyles DW, Burne TH, Reiss IK, Franco OH, Tiemeier H, Jaddoe VW, Duijts L. Associations of maternal and fetal 25-hydroxyvitamin D levels with childhood lung function and asthma: the Generation R Study. Clin Exp Allergy. 2016 Feb;46(2):337-46. doi: 10.1111/cea.12645. PMID 26399470
- [Background] Lange P, Celli B, Agusti A, Boje Jensen G, Divo M, Faner R, Guerra S, Marott JL, Martinez FD, Martinez-Camblor P, Meek P, Owen CA, Petersen H, Pinto-Plata V, Schnohr P, Sood A, Soriano JB, Tesfaigzi Y, Vestbo J. Lung-Function Trajectories Leading to Chronic Obstructive Pulmonary Disease. N Engl J Med. 2015 Jul 9;373(2):111-22. doi: 10.1056/NEJMoa1411532. PMID 26154786
- [Background] Postma DS, Bush A, van den Berge M. Risk factors and early origins of chronic obstructive pulmonary disease. Lancet. 2015 Mar 7;385(9971):899-909. doi: 10.1016/S0140-6736(14)60446-3. Epub 2014 Aug 11. PMID 25123778
- [Background] Belgrave DC, Buchan I, Bishop C, Lowe L, Simpson A, Custovic A. Trajectories of lung function during childhood. Am J Respir Crit Care Med. 2014 May 1;189(9):1101-9. doi: 10.1164/rccm.201309-1700OC. PMID 24606581
- [Result] Gonsard A, Marquant F, Elie C, Le Bourgeois M, Houdouin V, Delclaux C, Beydon N, Bellino A, Souberbielle JC, Sermet-Gaudelus I, Delacourt C, Benachi A, Hadchouel A. Specific airway resistance according to early maternal vitamin D status during pregnancy in children aged 5 to 6 years old from the FEPED cohort (RESPIFEPED). Eur J Pediatr. 2025 Feb 5;184(2):176. doi: 10.1007/s00431-024-05954-0. PMID 39907821